CLINICAL TRIAL: NCT04059094
Title: A Randomised, Double-blind, Placebo-controlled and Parallel Group Trial to Evaluate Efficacy and Safety of Twice Daily Inhaled Doses of BI 1265162 Delivered by Respimat® Inhaler as add-on Therapy to Standard of Care Over 4 Weeks in Patients With Cystic Fibrosis - BALANCE - CF™ 1
Brief Title: A 4-week Study to Test Different Doses of BI 1265162 in Adolescents and Adults With Cystic Fibrosis Using the Respimat® Inhaler - BALANCE - CF™1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not due to safety reasons
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1399-0003; 2019-000261-21 (EudraCT Number)
Record Dates: First submitted 2019-08-15; First posted 2019-08-16 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): 2 puffs ofmatching placebowere inhaledorally via theRespimat®inhaler twice dailyfor a treatmentperiod of 4 weeksin patients withcystic fibrosis.
  Interventions: Drug: Placebo
- BI 1265162 50 μg b.i.d. (Experimental): 2 puffs of 25micrograms (μg)BI 1265162(Total: 50μg)were inhaledorally via theRespimat®inhaler twice daily(b.i.d., daily dose:100μg) for atreatment periodof 4 weeks inpatients withcystic fibrosis.
  Interventions: Drug: BI 1265162
- BI 1265162 100 μg b.i.d. (Experimental): 2 puffs of 50micrograms (μg)BI 1265162(Total: 100μg)were inhaledorally via theRespimat®inhaler twice daily(b.i.d., daily dose:200μg) for atreatment periodof 4 weeks inpatients withcystic fibrosis.
  Interventions: Drug: BI 1265162
- BI 1265162 200 μg b.i.d. (Experimental): 2 puffs of 100micrograms (μg)BI 1265162(Total: 200μg)were inhaledorally via theRespimat®inhaler twice daily(b.i.d., daily dose:400μg) for atreatment periodof 4 weeks inpatients withcystic fibrosis.
  Interventions: Drug: BI 1265162
- BI 1265162 20 μg b.i.d. (Experimental): 2 puffs of 10micrograms (μg)BI 1265162(Total: 20μg)were inhaledorally via theRespimat®inhaler twice daily(b.i.d., daily dose:40μg) for atreatment periodof 4 weeks inpatients withcystic fibrosis.
  Interventions: Drug: BI 1265162

INTERVENTIONS:
Drug: BI 1265162 — Inhalation solution
  Arms: BI 1265162 100 μg b.i.d.; BI 1265162 20 μg b.i.d.; BI 1265162 200 μg b.i.d.; BI 1265162 50 μg b.i.d.
Drug: Placebo — Inhalation solution
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to assess the efficacy, safety and pharmacokinetics of twice daily inhaled doses of BI 1265162 delivered by Respimat® inhaler versus placebo in adolescents and adult patients with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 12 years of age or older at screening;
* Documented diagnosis of cystic fibrosis including:

  * positive sweat chloride ≥ 60 mEq/L, by pilocarpine iontophoresis OR
  * genotype with 2 identifiable mutations consistent with cystic fibrosis accompanied by one or more clinical features with cystic fibrosis phenotype;
* Patients able to perform acceptable spirometric manoeuvres according to American Thoracic Society (ATS) standards;
* FEV1 ≥ 40% and ≤ 90% of predicted values at screening and predose at Visit 2;
* Women of childbearing potential (WOCBP) must be willing and able to use highly effective methods of birth control per ICH M3 (R2) that result in a failure rate of less than1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient (or patient's legal guardian) information;
* Signed and dated written informed consent and assent in accordance with ICH Harmonized Guideline for Good Clinical Practice (GCP) and local legislation prior to admission in the trial.

Exclusion Criteria:

* Evidence of acute upper or lower respiratory tract infection within 4 weeks prior to randomization based on investigator's judgement;
* Pulmonary exacerbation requiring use of i.v./oral/inhaled antibiotics or oral corticosteroids within 4 weeks prior to randomisation;
* Patients with history of Acute Tubular Necrosis (ATN);
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix;
* Patients unable to inhale trial drug in an appropriate manner from the Respimat® inhaler based on investigator's judgement;
* Patients who have started a new chronic medication for CF within 4 weeks of randomisation;
* Patients who have previously received a lung transplant or patients who are currently on a waiting list to receive a lung transplant;
* Patients with a significant history of allergy/hypersensitivity (including medication allergy) which is deemed relevant to the trial as judged by the investigator or with a known hypersensitivity to trial drug or its components. "Significance" in this context refers to any increased risk of hypersensitivity reaction to trial medication;
* Any clinically significant laboratory abnormalities at screening as judged by the investigator, or any of the following:

  * Potassium > upper limit of normal (ULN) in non-haemolysed blood
  * Abnormal renal function defined as estimated Glomerular Filtration Rate (eGFR) < 60ml/min/1.73m²
  * Abnormal liver function, defined by serum level of either alanine transaminase (ALT), aspartate transaminase (AST) or total bilirubine ≥ 3 x upper limit of normal (ULN)
* Clinically significant disease or medical condition other than CF or CF-related conditions that, in the opinion of the investigator, would compromise the safety of the patient or the data quality. This includes significant haematological, hepatic, renal, cardiovascular and neurologic disease. Patients with diabetes may participate if their disease is under good control prior to screening;
* Patients not expected to comply with the protocol requirements or not expected to complete the trial as scheduled;
* Previous randomisation in this trial;
* Currently enrolled in another investigational device or drug trial, or less than 30 days or six half-lives (whichever is greater) since ending another investigational device or drug trial(s), or receiving other investigational treatment(s);
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable trial patient or unlikely to complete the trial;
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (8):
  - Nemours Children's Hospital, Orlando, Florida
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital of Pittsburgh of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University Health Systems, Richmond, Virginia
  - University of Washington, Seattle, Washington
- Belgium (2):
  - Brussels - UNIV UZ Brussel, Brussels
  - UZ Leuven, Leuven
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
- France (5):
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Robert Debré, Paris
  - HOP Cochin, Paris
  - HOP Lyon Sud, Pierre-Bénite
  - HOP Perharidy, Roscoff
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Universitätsklinikum Gießen und Marburg GmbH, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Tübingen, Tübingen
- Hospital Vall d'Hebron, Barcelona, Spain
- Sweden (2):
  - Sahlgrenska US, Göteborg, Gothenburg
  - Stockholm CF-Center , B59, Huddinge Universitetssjukhus, Stockholm
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https:// trials.boehringer-ingelheim.com/trial_results/ clinical_submission_documents.html to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link http://trials.boehringeringelheim. com/ to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://trials.boehringer-ingelheim.com

REFERENCES:
- [Derived] Goss CH, Fajac I, Jain R, Seibold W, Gupta A, Hsu MC, Sutharsan S, Davies JC, Mall MA. Efficacy and safety of inhaled ENaC inhibitor BI 1265162 in patients with cystic fibrosis: BALANCE-CF 1, a randomised, phase II study. Eur Respir J. 2022 Feb 17;59(2):2100746. doi: 10.1183/13993003.00746-2021. Print 2022 Feb. PMID 34385272
- [Derived] Goss CH, Jain R, Seibold W, Picard AC, Hsu MC, Gupta A, Fajac I. An innovative phase II trial to establish proof of efficacy and optimal dose of a new inhaled epithelial sodium channel inhibitor BI 1265162 in adults and adolescents with cystic fibrosis: BALANCE-CFTM 1. ERJ Open Res. 2020 Dec 7;6(4):00395-2020. doi: 10.1183/23120541.00395-2020. eCollection 2020 Oct. PMID 33313307
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial aimed to assess the efficacy, safety, and pharmacokinetics of different dose regimens of BI 1265162 taken twice daily by the Respimat® inhaler versus placebo in adult and adolescent patients with cystic fibrosis for a 4-week treatment period. Study was terminated without recruiting any adolescent patients.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo: 2 puffs of matching placebo were inhaled orally via the Respimat® inhaler twice daily for a treatment period of 4 weeks in patients with cystic fibrosis.
- BI 1265162 20μg b.i.d.: 2 puffs of 10 micrograms (μg) BI 1265162 (Total: 20μg) were inhaled orally via the Respimat® inhaler twice daily (b.i.d., daily dose: 40μg) for a treatment period of 4 weeks in patients with cystic fibrosis.
- BI 1265162 50μg b.i.d.: 2 puffs of 25 micrograms (μg) BI 1265162 (Total: 50μg) were inhaled orally via the Respimat® inhaler twice daily (b.i.d., daily dose: 100μg) for a treatment period of 4 weeks in patients with cystic fibrosis.
- BI 1265162 100μg b.i.d.: 2 puffs of 50 micrograms (μg) BI 1265162 (Total: 100μg) were inhaled orally via the Respimat® inhaler twice daily (b.i.d., daily dose: 200μg) for a treatment period of 4 weeks in patients with cystic fibrosis.
- BI 1265162 200μg b.i.d.: 2 puffs of 100 micrograms (μg) BI 1265162 (Total: 200μg) were inhaled orally via the Respimat® inhaler twice daily (b.i.d., daily dose: 400μg) for a treatment period of 4 weeks in patients with cystic fibrosis.
Period: Overall Study
Arm/Group | Placebo | BI 1265162 20μg b.i.d. | BI 1265162 50μg b.i.d. | BI 1265162 100μg b.i.d. | BI 1265162 200μg b.i.d.
Started | 18 | 6 | 5 | 5 | 18
Completed | 18 | 4 | 5 | 5 | 17
Not Completed | 0 | 2 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Not willing to travel due to COVID-19 pandemic | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all patients who were randomized and treated with at least one dose of study drug. The treatment assignment was determined based on the first treatment the subjects received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 1265162 20μg b.i.d. | BI 1265162 50μg b.i.d. | BI 1265162 100μg b.i.d. | BI 1265162 200μg b.i.d. | Total
Number analyzed (Participants) | 18 | 6 | 5 | 5 | 18 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.3 (10.1) | 26.8 (5.8) | 31.2 (8.6) | 36.8 (4.2) | 33.4 (10.2) | 31.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 1 | 3 | 10
  Male | 16 | 5 | 2 | 4 | 15 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 17 | 6 | 5 | 5 | 18 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 17 | 6 | 5 | 4 | 18 | 50
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Trough forced expiratory volume in one second (FEV1) percent predicted [Mean (Standard Deviation); unit: Percentage of predicted trough FEV1] — Baseline trough FEV1 percent (%) predicted was defined as the last measurement taken on day 1 before first study drug administration and was measured within 30 minutes prior to dosing. Population: Treated set (TS): The TS included all patients who were randomized and treated with at least one dose of study drug. The treatment assignment was determined based on the first treatment the subjects received. One participant in the BI 1265162 200 microgram group did not have valid baseline trough FEV1 percent predicted value measured.
  Percentage of predicted trough FEV1
    number analyzed (Participants) | 18 | 6 | 5 | 5 | 17 | 51
    (all) | 59.40 (11.29) | 69.93 (15.99) | 63.02 (14.40) | 65.50 (7.00) | 57.94 (13.76) | 61.11 (12.89)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent Predicted Trough Forced Expiratory Volume in 1 Second (FEV1) After 4 Weeks of Treatment
Description: Trough FEV1 was measured within 30 minutes prior to dosing of study medication.
Time Frame: At 30 minutes prior to dosing in Day 1 (baseline) and Day 29 (end of 4-week treatment period).
Population: Treated set (TS): The TS included all patients who were randomized and treated with at least one dose of study drug. The treatment assignment was determined based on the first treatment the subjects received. Only participants with non-missing outcome measured were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of predicted trough FEV1
Arm/Group | Placebo | BI 1265162 20μg b.i.d. | BI 1265162 50μg b.i.d. | BI 1265162 100μg b.i.d. | BI 1265162 200μg b.i.d.
Number analyzed (Participants) | 17 | 4 | 5 | 5 | 16
Percentage of predicted trough FEV1 | -0.6 (8.03) | -0.5 (2.82) | -0.22 (2.62) | 2.82 (3.57) | 0.45 (5.42)
Statistical Analysis 1: Comparison: Placebo vs BI 1265162 200μg b.i.d; Mixed Model for Repeated Measures (MMRM) with fixed effects for baseline, visit, treatment, treatment-by-visit interaction, baseline-by-visit interaction, and random effect for patient was applied. No hypothesis testing was performed, as this trial was prematurely discontinued. MMRM only included data from 200µg BI and placebo, as the sample size of the BI 20µg, BI 50µg and BI 100µg dose levels was limited because of the premature discontinuation of the trial; Test type: Other; p = 0.5468, Mixed model with repeated measurements; Adjusted means difference = 1.5, 95% CI 2-sided [-3.5 to 6.5], Standard Error of Mean 2.45 — Adjusted means difference was calculated as value from BI 1265162 200μg minus value from placebo group

2. Secondary Outcome: Change From Baseline in Lung Clearance Index (LCI) Assessed by N2 Multiple Breath Washout (N2MBW) Procedure After 4 Weeks of Treatment
Description: Change from baseline in Lung Clearance Index (LCI) assessed by N2 Multiple Breath Washout (N2MBW) procedure after 4 weeks of treatment was reported. LCI was calculated as the ratio of cumulative expired volume (CEV) to functional residual capacity (FRC), which was LCI = CEV (milliliter/kilogram) / FRC (milliliter/kilogram) and hence, LCI was "Unitless". The change from baseline after 4 weeks of treatment in LCI was then calculated as the LCI value measured after 4 weeks of treatment at Day 29 minus the LCI value measured at baseline on Day 1.
Time Frame: At pre-dose in Day 1 (baseline) and Day 29 (end of 4-week treatment period).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Placebo | BI 1265162 20μg b.i.d. | BI 1265162 50μg b.i.d. | BI 1265162 100μg b.i.d. | BI 1265162 200μg b.i.d.
Number analyzed (Participants) | 6 | 0 | 1 | 1 | 3
Unitless | -0.824 (3.312) |  | -0.238 (NA) — Data from only one patients was available and no standard deviation could be calculated. | -2.547 (NA) — Data from only one patients was available and no standard deviation could be calculated. | -0.081 (1.001)
Statistical Analysis 1: Comparison: Placebo vs BI 1265162 200μg b.i.d; ANCOVA based on analysis of covariance with fixed effects for baseline and treatment was applied. Statistical analysis was performed for 200μg BI and placebo groups only. No hypothesis testing was performed, as this trial was prematurely discontinued. ANCOVA only included data from 200µg BI and placebo, as the sample size of the BI 20µg, BI 50µg and BI 100µg dose levels was limited because of the premature discontinuation of the trial; Test type: Other; p = 0.3039, ANCOVA; Adjuste means difference = 2.1, 95% CI 2-sided [-2.4 to 6.5], Standard Error of Mean 1.83 — Adjusted means difference was calculated as value from BI 1265162 200μg minus value from placebo group

3. Secondary Outcome: Change From Baseline in Cystic Fibrosis Questionnaire Revised (CFQ-R) Total Score After 4 Weeks of Treatment
Description: The adult/adolescent format of the CFQ-R consists of 50 questions (qts) dividing into 12 domains: Physical functioning(8 qts), role limitations(4 qts), vitality(4 qts), emotional functioning(5 qts), social functioning(6 qts), body image(3 qts), eating disturbance(3 qts), treatment burden(3 qts), health perceptions(3 qts), weight(1 qts), respiratory symptoms(7 qts), and digestive system(3 qts). The score of some qts is first reversed if reversed coded, so that the score for each of the 50 qts ranges from 1 to 4 points (less symptoms). Then, a domain score for a domain with N qts is calculated as (sum of the scores of the N qts - N)/(N ✕ 4 - N) ✕ 100. Each domain score ranges from 0 to 100 (better health). The CFQ-R total score is summing up the domain scores and ranges from 0 to 1200 (better quality of life). The change from baseline in Cystic Fibrosis Questionnaire Revised (CFQ-R) total score after 4 weeks of treatment was reported.
Time Frame: At Day 1 (baseline) and Day 29 (end of 4-week treatment period).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | BI 1265162 20μg b.i.d. | BI 1265162 50μg b.i.d. | BI 1265162 100μg b.i.d. | BI 1265162 200μg b.i.d.
Number analyzed (Participants) | 18 | 6 | 5 | 5 | 16
Score on a scale | 5.941 (76.669) | 27.083 (61.626) | 11.167 (33.968) | -15.611 (62.167) | 24.236 (58.290)

4. Secondary Outcome: Change From Baseline in Cough and Sputum Assessment Questionnaire (CASA-Q) (4 Separate Sub-scores) After 4 Weeks of Treatment
Description: The 20-item Sputum Assessment Questionnaire (CASA-Q) consisted of 4 domains: Cough Symptoms Domain (3 items), Cough Impact Domain (8 items), Sputum Symptoms Domain (3 items), and Sputum Impact Domain (6 items). Score of each item has been reversed such that better responses have higher score, which ranges from 1 (worse) to 5 (better health). For each domain, the domain score was calculated by summing up the scores of the respective items and scaling to a value ranging from 0 to 100, with higher score associated with fewer symptoms/less impact due to cough or sputum. The 4 domain scores (sub-scores) were reported.
Time Frame: At Day 1 (baseline) and Day 29 (end of 4-week treatment period).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | BI 1265162 20μg b.i.d. | BI 1265162 50μg b.i.d. | BI 1265162 100μg b.i.d. | BI 1265162 200μg b.i.d.
Number analyzed (Participants) | 18 | 4 | 5 | 5 | 17
Score on a scale
  Cough Symptom Domain Score | 4.167 (18.798) | 10.417 (17.180) | 8.333 (8.333) | 3.333 (24.008) | 5.392 (15.574)
  Cough Impact Domain Score | -0.521 (16.648) | -6.250 (12.758) | -0.625 (12.771) | 1.250 (14.757) | 0.735 (11.187)
  Sputum Symptom Domain Score | 5.093 (15.950) | 4.167 (8.333) | 10.000 (14.907) | 3.333 (16.245) | 5.392 (19.530)
  Sputum Impact Domain Score | -0.694 (16.497) | -4.167 (3.402) | 5.000 (11.562) | -0.833 (13.944) | 0.490 (11.110)

5. Secondary Outcome: Percentage of Patients With Treatment-emergent Adverse Events (AE) up to Day 36
Description: Percentage of patients with any treatment-emergent Adverse Events (AE) up to day 36 was reported.
Time Frame: From Day 1 (baseline) until end of 4 weeks of treatment period (Day 29) plus 7 days of follow-up, up to 36 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | BI 1265162 20μg b.i.d. | BI 1265162 50μg b.i.d. | BI 1265162 100μg b.i.d. | BI 1265162 200μg b.i.d.
Number analyzed (Participants) | 18 | 6 | 5 | 5 | 18
Percentage of participants | 66.7 | 0 | 40.0 | 40.0 | 83.3

6. Secondary Outcome: Concentration of BI 1265162 in Plasma at 0.083 Hour at Steady State Following Dose 15 (C0.083,ss,15)
Description: Concentration of BI 1265162 in plasma at 0.083 hour at steady state following dose 15 (C0.083,ss,15) was reported.
Time Frame: At 5 minutes (around 0.083 hours) post dosing at steady state on Day 8 for dose 15 (morning dose on Day 8).
Population: Pharmacokinetic set (PKS): The PKS included all patients in the treated set who provided at least one pharmacokinetic parameter. Only participants with non-missing outcome measured were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole/liter (pmol/L)
Arm/Group | BI 1265162 20μg b.i.d. | BI 1265162 50μg b.i.d. | BI 1265162 100μg b.i.d. | BI 1265162 200μg b.i.d.
Number analyzed (Participants) | 3 | 4 | 4 | 16
picomole/liter (pmol/L) | 207 (59.9) | 471 (30.0) | 1010 (20.1) | 1110 (84.8)

7. Secondary Outcome: Concentration of BI 1265162 in Plasma at 0.083 Hour at Steady State Following Dose 57 (C0.083,ss,57)
Description: Concentration of BI 1265162 in plasma at 0.083 hour at steady state following dose 57 (C0.083,ss,57) was reported.
Time Frame: At 5 minutes (around 0.083 hours) post dosing at steady state on Day 29 for dose 57 (morning dose on Day 29).
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole/liter (pmol/L)
Arm/Group | BI 1265162 20μg b.i.d. | BI 1265162 50μg b.i.d. | BI 1265162 100μg b.i.d. | BI 1265162 200μg b.i.d.
Number analyzed (Participants) | 3 | 3 | 5 | 14
picomole/liter (pmol/L) | 162 (76.3) | 463 (15.4) | 573 (94.0) | 1080 (165)

8. Secondary Outcome: Pre-dose Concentration Measured of BI 1265162 in Plasma at Steady State After Dose 15 (Cpre,ss, 15)
Description: Pre-dose concentration measured of BI 1265162 in plasma at steady state after dose 15 (Cpre,ss, 15) was reported.
Time Frame: At pre-dose (taken within 60 minutes prior to dosing) at steady state on Day 8 for dose 15 (morning dose on Day 8).
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole/liter (pmol/L)
Arm/Group | BI 1265162 20μg b.i.d. | BI 1265162 50μg b.i.d. | BI 1265162 100μg b.i.d. | BI 1265162 200μg b.i.d.
Number analyzed (Participants) | 3 | 4 | 5 | 14
picomole/liter (pmol/L) | 7.82 (28.0) | 24.3 (31.8) | 38.4 (292) | 43.8 (95.6)

9. Secondary Outcome: Pre-dose Concentration Measured of BI 1265162 in Plasma at Steady State After Dose 57 (Cpre,ss, 57)
Description: Pre-dose concentration measured of BI 1265162 in plasma at steady state after dose 57 (Cpre,ss, 57) was reported.
Time Frame: At pre-dose (taken within 60 minutes prior to dosing) at steady state on Day 29 for dose 57 (morning dose on Day 29).
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole/liter (pmol/L)
Arm/Group | BI 1265162 20μg b.i.d. | BI 1265162 50μg b.i.d. | BI 1265162 100μg b.i.d. | BI 1265162 200μg b.i.d.
Number analyzed (Participants) | 1 | 3 | 3 | 12
picomole/liter (pmol/L) | NA (NA) — No descriptive statistics calculated since not enough data as only 1 patient was analyzed. | 13.0 (80.8) | 22.3 (48.3) | 37.2 (56.9)

10. Secondary Outcome: Area Under the Concentration-time Curve of BI 1265162 in Plasma From 0 to 4 Hours at Steady State After Dose 15 (AUC0-4,ss,15)
Description: Area under the concentration-time curve of BI 1265162 in plasma from 0 to 4 hours at steady state after dose 15 (AUC0-4,ss,15) was reported.
Time Frame: At pre-dose (taken within 60 minutes prior to dosing) and 5 minutes (min), 30 min, 1 hour, and 4 hours post dosing at steady state on Day 8 for dose 15 (morning dose on Day 8).
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * picomole/liter (h*pmol/L)
Arm/Group | BI 1265162 20μg b.i.d. | BI 1265162 50μg b.i.d. | BI 1265162 100μg b.i.d. | BI 1265162 200μg b.i.d.
Number analyzed (Participants) | 5 | 4 | 4 | 17
hours * picomole/liter (h*pmol/L) | 192 (45.3) | 541 (19.1) | 1020 (8.93) | 1380 (71.0)

ADVERSE EVENTS:
Time Frame: From Day 1 (baseline) until end of 4 weeks of treatment period (Day 29) plus 7 days of follow-up, up to 36 days.
Description: Treated set (TS): The TS included all patients who were randomized and treated with at least one dose of study drug. The treatment assignment was determined based on the first treatment the subjects received.
Arm/Group | Placebo | BI 1265162 20μg b.i.d. | BI 1265162 50μg b.i.d. | BI 1265162 100μg b.i.d. | BI 1265162 200μg b.i.d.
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/6 | 0/5 | 0/5 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/6 | 0/5 | 0/5 | 1/18
Other Adverse Events (participants affected / at risk) | 11/18 | 0/6 | 2/5 | 2/5 | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | BI 1265162 20μg b.i.d. (N=6) | BI 1265162 50μg b.i.d. (N=5) | BI 1265162 100μg b.i.d. (N=5) | BI 1265162 200μg b.i.d. (N=18)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | BI 1265162 20μg b.i.d. (N=6) | BI 1265162 50μg b.i.d. (N=5) | BI 1265162 100μg b.i.d. (N=5) | BI 1265162 200μg b.i.d. (N=18)
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 0 | 0 | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Pulmonary function test decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This trial was prematurely discontinued with only adult patients being recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT04059094/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT04059094/SAP_001.pdf